CLINICAL TRIAL: NCT06704360
Title: A Single-blind Randomized Controlled Trial to Evaluate Efficacy and Safety of Immersive Virtual Reality for Post-stroke Cognitive Impairment
Brief Title: Efficacy and Safety of Immersive Virtual Reality for Post-stroke Cognitive Impairment
Acronym: EVRPSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dingqun Bai (Other)
Responsible Party: Sponsor-Investigator, Dingqun Bai, Director of rehabilitation Medicine, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241120
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Cognitive Decline
Keywords: stroke; virtual reality; fNIRS; cognitive impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (virtual reality cognitive training group) (Experimental): Immersive VR cognitive training with suitable training intensity.
  Interventions: Device: immersive VR pathfinding training
- OT group (occupational therapy group) (Active Comparator): Conventional cognitive training (occupational therapy) with suitable training intensity.
  Interventions: Other: Occupational therapy

INTERVENTIONS:
Device: immersive VR pathfinding training — Pathfinding training with immersive VR.
  Arms: VR group (virtual reality cognitive training group)
Other: Occupational therapy — Only receive conventional cognitive training group
  Arms: OT group (occupational therapy group)

SUMMARY:
This is a single-blind randomized controlled trial to evaluate the efficacy and safety of immersive virtual reality for post-stroke cognitive impairment.

DETAILED DESCRIPTION:
This is a single-blind randomized controlled intervention study. Each stroke subject will undergo screening period, baseline assessment period, intervention period, endpoint assessment period.

In the screening period, the verification of inclusion/exclusion criteria and the acquisition of informed consent will be completed.

In the baseline assessment period and endpoint assessment period, cognitive function related scale assessment included Mental State Examination Scale (MMSE), Montreal Cognitive Assessment (MoCA), drawing clock test (DCT), Shape trials test A.B (STT-A, STT-B), standardized digital modal test (SDMT), auditory verbal learning test-Huashan version (AVLT-H), and activity of daily living (ADL) scale will be used to evaluate the function of each patient. Meanwhile, brain functional activation of each patient during the cognitive task (Stroop task, 1-back task and verbal fluency test) will be evaluated using functional near-infrared spectroscopy (fNIRS).

In the intervention period, the VR group will receive immersive VR cognitive training with suitable for training intensity and the control group will receive the conventional cognitive train (occupational therapy) with suitable for training intensity in the control group. The training will lasted 20 minutes per time, 5 times per week for four weeks, with a total of 600 minutes, training frequency will be adjusted according to the patient's own conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke by neuroimaging (CT or MRI) assessment
2. 18-85 years old
3. Be able to follow instructions to complete the test
4. Can tolerate the rehabilitation training of this experiment
5. First stroke
6. Patients who signed informed consent

Exclusion Criteria:

1. The test could not be tolerated due to organic disease
2. There is a serious mental illness resulting in inability to cooperate with or tolerate this test
3. is participating in another clinical trial involving an investigational drug or physical therapy
4. Patients who have not signed informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mental State Examination Scale (MMSE) | 1. finished in 3 days before training. 2. finished 3 days after 30-days training
  Global cognitive function assessment. Easy to use and one of the most used scales to screen person with cognitive impairment in the world. The minimum and maximum values range from 0 to 30. Higher score means better cognition level.
Montreal Cognitive Assessment (MoCA) | 1. finished in 3 days before training. 2. finished 3 days after 30-days training
  one of the most used scales to assess cognition and screen person with cognitive impairment in the world. The minimum and maximum values range from 0 to 30. Higher score means better cognition level.
Brain functional activation (fNIRS) | 1. finished in 3 days before training. 2. finished 3 days after 30-days training
  Brain functional activation of each patient during the cognitive task (Stroop task, 1-back task and verbal fluency test) will be evaluated using functional near-infrared spectroscopy (fNIRS).

CONTACTS AND LOCATIONS:
Overall Officials: Dingqun Bai, Study Chair — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: Undecided